CLINICAL TRIAL: NCT01854086
Title: Compliance and Persistence With Osteoporosis Treatment and Attitude Towards Future Therapy Among Post-menopausal Israeli Women During Drug Treatment or Drug Holiday: Data From a Single Outpatient Endocrine Clinic.
Brief Title: Compliance and Persistence With Osteoporosis Treatment and Attitude Towards Future Therapy Among Post-menopausal Israeli Women During Drug Treatment or Drug Holiday
Acronym: CONTINUITY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC130009-13CTIL
Record Dates: First submitted 2013-05-06; First posted 2013-05-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Osteoporosis
Keywords: osteoporosis; postmenopausal; patient compliance; compliance; diphosphonates; bisphosphonates
MeSH Terms: conditions — Osteoporosis; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postmenopausal women: Postmenopausal women treated with bisphosphonates
  Interventions: Other: Questionnaires about compliance and persistence with bisphosphonates treatment

INTERVENTIONS:
Other: Questionnaires about compliance and persistence with bisphosphonates treatment

SUMMARY:
The purpose of the study is to provide information about the rate of response and persistence to drug therapies for osteoporosis. Another issue examined in this study refers to the preferences and concerns about future treatments in patients during "drug holiday".

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Diagnosis of osteoporosis in the medical record
* At least one prescription drug to treat osteoporosis in the last 5 years
* Insured by "Clalit" Health Services
* Hebrew-speaking capability and readiness to answer a questionnaire

Exclusion Criteria:

* Premenopausal women
* No diagnosis of osteoporosis in the medical record
* No treatment for osteoporosis in the last 5 years
* Women who do not speak Hebrew or are unable to answer a questionnaire

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with osteoporosis,who been treated in Endocrinology Clinic of Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Compliance and persistence to osteoporosis drug therapy | Participants will be followed for the duration of their clinic visit, an average of 5 hours
  Data collection will be done by questionnaires and from the medical record of the patient. The information collected will include: demographic information, measurements of bone density, additional information about the disease and treatment that the patient receives,prescription purchases and additional drugs the patient is taking (steroids, PPI's(Proton Pump Inhibitors) / H2 receptor antagonists and NSAIDs(Non Steroidal Anti Inflammatories)).

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center the clalit health care services group, Kfar Saba, Israel

REFERENCES:
- [Result] Cramer JA, Amonkar MM, Hebborn A, Altman R. Compliance and persistence with bisphosphonate dosing regimens among women with postmenopausal osteoporosis. Curr Med Res Opin. 2005 Sep;21(9):1453-60. doi: 10.1185/030079905X61875. PMID 16197664